CLINICAL TRIAL: NCT06331572
Title: Exploring Blood Plasma Metabolomics: Unraveling the Metabolic Landscape in Treatment-Resistant Adolescent Depression
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Zhou, professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 1stChongqingMU-TRD
Record Dates: First submitted 2024-03-20; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Psychiatric Disorder; Major Depressive Disorder; Metabolic Disorder
Keywords: adolescent MDD; treatment-resistant depression; metabolomic
MeSH Terms: conditions — Mental Disorders; Depressive Disorder, Major; Metabolic Diseases; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Staging of diseases in the inclusion exclusion criteria refer to previous studies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- TRD: 1. age 12-18 years
  2. Meet the diagnostic criteria for MDD according to the DSM-5
  3. HAMD-17 score > 13
  4. currently or previously taking a standard therapeutic dose of antidepressant for at least 6 weeks, and they had at least one historical failure to an antidepressant (reduction in depressive symptoms <50%)
  Interventions: Diagnostic Test: 17-HAMD
- FEDN-MDD: 1. age 12-18 years 2. Meet the diagnostic criteria for MDD according to the DSM-5 2. First-episode and drug-naive 4. HAMD-17 score > 17
  Interventions: Diagnostic Test: 17-HAMD
- HC: 1. age 12-18 years
  2. HAMD-17 score < 7
  3. HCs without a personal history of a mental illness or family history in a first-degree relative
  Interventions: Diagnostic Test: 17-HAMD

INTERVENTIONS:
Diagnostic Test: 17-HAMD — Patients were interviewed in a semi-structured manner and assessed using the 17-item Hamilton Depression Scale and the Hamilton Anxiety Scale
  Other Names: HAMA

SUMMARY:
This study contributes new evidence for the identification of adolescent TRD and sheds light on differing pathophysiologies by delineating distinct plasma metabolic profiles between adolescent TRD and FEDN-MDD.

ELIGIBILITY:
Inclusion Criteria:

FEDN-MDD：

1. Age 12-18 years
2. Meet the diagnostic criteria for MDD according to the DSM-5
3. First-episode and drug-naive
4. HAMD-17 score > 17

TRD:

1. Age 12-18 years
2. Meet the diagnostic criteria for MDD according to the DSM-5
3. HAMD-17 score > 13
4. Currently or previously taking a standard therapeutic dose of antidepressant for at least 6 weeks, and they had at least one historical failure to an antidepressant (reduction in depressive symptoms <50%)

HC:

1. age 12-18 years
2. HAMD-17 score < 7
3. HCs without a personal history of a mental illness or family history in a first-degree relative

Exclusion Criteria:

FEDN-MDD、TRD：

1. the presence or past history of severe medical, neurological or psychiatric disorders (other than MDD in patients)
2. anxiety comorbidity was not considered an exclusion criterion provided that MDD was the main diagnosis and the primary reason for seeking assistance
3. substance abuse, head trauma, or loss of consciousness
4. Chronic physical diseases that significantly affect peripheral metabolism or neurological function
5. Pregnant and lactating women

HC:

1. the presence or past history of severe medical, neurological or psychiatric disorders
2. substance abuse, head trauma, or loss of consciousness
3. Chronic physical diseases that significantly affect peripheral metabolism or neurological function
4. Pregnant and lactating women

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: FEDN-MDD: 53 patients with MDD who had a first episode and had not been treated with antidepressants TRD: 53 patients who had been on medication for at least 6 weeks or more and were not responding to antidepressant therapy HC: 56 healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
17 items Hamilton Depression Scale | baseline
  The Hamilton Depression Scale assesses the level of depressive symptoms in patients

SECONDARY OUTCOMES:
Hamilton Anxiety Scale | baseline
  The Hamilton Anxiety Scale assesses the level of anxiety symptoms in patients

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Province, China